CLINICAL TRIAL: NCT07002801
Title: Application of Remimazolam Combined With Esketamine in Painless Gastroscopy and Colonoscopy in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Shi xiaoqian, Graduate student, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChiCTR2500098650
Record Dates: First submitted 2025-05-12; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Disease
Keywords: remimazolam; esketamine; painless gastroscopy and colonoscopy; success rate of calming down
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the anesthesiologist nor the operator of the gastroscopy was aware of it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remimazolam plus esketamine group (Experimental): Esketamine combined with remimazolamwas used for anesthesia.
  Interventions: Combination Product: remimazolam-esketamine
- remimazolam plus remifentanil group (Active Comparator): Remifentanil combined with remimazolam was used for anesthesia.
  Interventions: Combination Product: remimazolam-remifentanil

INTERVENTIONS:
Combination Product: remimazolam-remifentanil — For elderly patients scheduled for elective painless gastro-intestinal endoscopy, remimazolam 0.2mg/kg and remifentanil 0.2ug/kg are used for anesthesia induction. During the operation, the doses are adjusted according to the depth of sedation of the patients.
  Arms: remimazolam plus remifentanil group
Combination Product: remimazolam-esketamine — For elderly patients scheduled for painless gastroenterological endoscopy, remimazolam 0.2mg/kg and esketamine 0.15mg/kg are used for anesthesia induction. During the operation, the dosage is adjusted according to the patient's level of sedation.
  Arms: remimazolam plus esketamine group

SUMMARY:
The objective of this clinical trial is to assess the feasibility of the remimazolam combined with esketamine OFA (opioid-free anesthesia) protocol for painless gastroscopy and colonoscopy in elderly patients and to determine if it is non-inferior to the traditional OA (opioid-containing anesthesia) protocol. The main questions it aims to answer are:

* Is the remimazolam combined with esketamine protocol feasible for painless gastroscopy and colonoscopy in elderly patients?
* Is the OFA protocol superior to the OA protocol?

Participants will:

* During anesthesia induction, the experimental group will receive remimazolam combined with esketamine for anesthesia, while the control group will receive remimazolam combined with remifentanil.
* Record respiratory and circulatory indicators and adverse reaction times.

DETAILED DESCRIPTION:
Elderly patients undergoing painless gastroenteroscopy were randomly divided into remazolam + esketamine group (RE group) and remazolam + remifentanil group (RR group). In RE group, anesthesia induction was as follows: Remazolam 0.2mg/kg, esketamine 0.15mg/kg, lidocaine 0.5mg/kg, changtonine 0.2mg. RR group: Anesthesia induction: remazolam 0.2mg/kg, remifentanil 0.2μg/kg, lidocaine 0.5mg/kg, Changtonine 0.2mg. Remazolam and esketamine/remifentanil were added during the operation according to the depth of sedation and movement of the patient. The outcome measures included success rate of sedation, incidence of respiratory depression, incidence of hypotension and bradycardia, postoperative recovery time, incidence of adverse reactions, postoperative satisfaction of patients and gastroenteroscopists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing painless gastroenteroscopy in outpatient clinics;
2. aged 65 years and above;
3. American Society of Anesthesiologists (ASA) grades I - III.

Exclusion Criteria:

1. Patients with abnormal liver or kidney function;
2. known respiratory or endocrine diseases;
3. Patients with uncontrolled hypertension and NYHA classification Ⅲ-Ⅳ;
4. Taking monoamine oxidase inhibitors, sedatives, analgesics, hypnotics, antipsychotics, antiemetics or antidepressants;
5. Addiction to tobacco and alcohol;
6. Patients allergic to the investigational drug;
7. expected difficult airway;
8. Body mass index (BMI) >35kg/m^2;
9. Have participated in other clinical trials within the past three months;
10. Patients with psychosocial illness or cognitive dysfunction and inability to cooperate or communicate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Sedation success rate | From the start of anesthesia induction to the end of the surgery
  Successful sedation：① The patient underwent painless gastroenteroscopy;②During anesthesia induction, a single remazolam is not enough to achieve sufficient sedation depth, and it needs to be remedied, and the number of remediations within 15min is less than 5 times; Intraoperative supplementary times ≤5 times within any 15min.③ The patient did not use rescue drugs;Sedation success rate: Number of patients successfully sedated/total number of patients included in the data analysis for this group
Incidence of hypotension | From the start of anesthesia induction to the end of the surgery
  Hypotension: systolic blood pressure below 80% of baseline systolic blood pressure or MAP below 80% of baseline MAP; Incidence of hypotension: Number of patients with intraoperative hypotension/total number of patients included in the data analysis for this group

SECONDARY OUTCOMES:
degree of blood oxygen saturation | From the start of anesthesia induction to the end of the surgery
  The blood oxygen saturation was recorded every 2 minutes during the operation. The maximum value is 100. An event where blood oxygen saturation drops below 90 is described as respiratory depression.
respiratory rate | From the start of anesthesia induction to the end of the surgery
  The respiratory rate was recorded every 2 minutes during the operation. The normal breathing rate is 12 to 20 breaths per minute.
bispectral index | From the start of anesthesia induction to the end of the surgery
  During the surgery, the bilateral frequency index of brain electricity was recorded every 2 minutes. The bispectral index of electroencephalogram is mainly used to assess the depth of sedation, the effect of anesthesia and the state of consciousness. Its value range is from 0 to 100. The higher the value, the higher the degree of consciousness; the lower the value, the deeper the degree of brain inhibition.
Heart rate | From the start of anesthesia induction to the end of the surgery
  The heart rate was recorded every 2 minutes during the operation. The normal heart rate is 60 to 100 beats per minute.
Blood pressure | From the start of anesthesia induction to the end of the surgery
  The blood pressure was recorded every 2 minutes during the operation.
Modified Observer's Assessment of Alertness/Sedation Scale | From the start of anesthesia induction to the end of the surgery
  The MOAA/S, which stands for Modified Observer's Assessment of Alertness/Sedation Scale, assesses the patient's response to sounds or physical stimuli and is scored on a scale of 6 levels:
  Level 5: Normal alertness, quick response to normal tone of voice; Level 4: Slow response to normal tone of voice; Level 3: Only responds to loud or repeated calls; Level 2: Only responds to slight shaking or tactile stimuli; Level 1: No response to slight shaking or tactile stimuli, but responds to pain stimuli (such as pinching the trapezius muscle); Level 0: No response to pain stimuli. During the surgery, the MOAA/S value was recorded every 2 minutes.
Hiccup | From the start of anesthesia induction to the end of the surgery
  Level 0: No hiccups; Level 1: Single mild hiccup; Level 2: Multiple mild hiccups, not affecting the surgical operation (≤ 5 seconds); Level 3: Severe hiccups, affecting the surgical operation (> 5 seconds).
cough | From the start of anesthesia induction to the end of the surgery
  Level 0: No choking coughing action; Level 1: A single mild choking coughing action; Level 2: Multiple mild choking coughing actions, which do not affect the surgical operation (≤ 5 seconds); Level 3: Severe coughing (> 5 seconds).
Physical movement | From the start of anesthesia induction to the end of the surgery
  Level 1: No activity: Level 2: Slight activity, does not affect operation: Level 3: Obvious activity, has some impact on surgical operation; Level 4: Limb twisting, significantly affects operation.
Grade of abdominal wall muscle stiffness | From the start of anesthesia induction to the end of the surgery
  No; moderate (by pressing the abdomen, the abdominal wall muscles become stiff, which affects the colonoscopy examination); Severe (by pressing the abdomen, the abdominal wall muscles become stiff, severely affecting the colonoscopy examination)
time index | From the start of anesthesia induction to the end of the surgery
  The induction time of anesthesia is the period from the start of administering remimazolam and remifentanil (esketamine) until the patient loses consciousness and is ready for surgery. The operation time is the duration from the beginning of the gastroscopy procedure to the end of the colonoscopy. The period of full consciousness is from the last administration of anesthetic drugs until the patient regains consciousness. The anesthesia recovery time is the duration from the time the patient regains consciousness to the time when the Aldrete score reaches 9 points.
The usage of anesthetic drugs | From the start of anesthesia induction to the end of the surgery
  Record the consumption amounts of lidocaine, esketamine, remifentanil and remimazolam during the operation
Adverse event | From the induction of anesthesia to the end of the surgery, and from the end of the surgery to the time when the patient leaves the anesthesia recovery room.
  Adverse events include intraoperative respiratory depression, hypotension, hypertension, bradycardia, tachycardia, arrhythmia, hiccups, choking cough, body movement, abdominal wall rigidity; postoperative nausea, vomiting, headache, dizziness, visual impairment, hallucination, intraoperative awareness, etc.
The satisfaction of patients | Ask the patient after they regain consciousness.
  The patient's satisfaction was measured using the visual analogue scale method. A 10-cm movable ruler with 10 marks was used, with the two ends marked as 0 and 10 respectively. The patient was asked to mark the corresponding position on the ruler that represented their satisfaction level. 0 represented extreme dissatisfaction and 10 represented very satisfaction.
The satisfaction of doctor | At the end of the surgery
  The satisfaction of the doctors was measured using the visual analogue scale method. A 10-cm movable ruler was used, marked with 10 graduations, with the two ends representing 0 points and 10 points respectively. The doctors were asked to mark the corresponding position on the ruler that best represented their satisfaction level. 0 points indicated extreme dissatisfaction, while 10 points indicated very high satisfaction.
Patient pain score | After the patient regained consciousness
  The patient's pain score is classified into four levels: no pain, mild abdominal distension pain (pain is present only when pressed; no pain when not pressed), moderate abdominal pain (pain persists even when not pressed, but is tolerable), and severe abdominal pain (pain is unbearable).
Telephone Interview for Cognitive Status | Before the start of the surgery, after the anesthesia wore off, and on the seventh day after the surgery
  The Telephone Interview for Cognitive Status is a tool used to assess cognitive functions, especially suitable for remote screening of cognitive impairments. TICS is a standardized telephone interview scale that evaluates the cognitive functions of the subjects through questions, including orientation, memory, language ability, calculation ability, etc. It consists of 13 items, with a total score ranging from 0 to 50, and a lower score indicates more severe cognitive impairment.
The Confusion Assessment Method---CAM | The seventh day after the operation
  1. Applicable population: Elderly patients, especially those who have undergone surgery or have cognitive impairments.
  2. Assessment items: It includes 11 indicators, such as acute onset, attention disorder, disordered thinking, disorientation, etc. Each item is scored from 0 to 3 or 0 to 4 points.
  3. Diagnostic criteria: Total score: Below 19 points indicates no delirium, 20 to 22 points indicates suspicion, and above 22 points confirms the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: SHI Jinghui SHI, Study Director
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Yes
The original data sharing platform (IPD sharing platform) of ResMan, a clinical trial registration center of China, on June 30, 2028.
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: http://www.medresman.org.cn/pub/cn/help.aspx